CLINICAL TRIAL: NCT03425149
Title: A Randomized, Placebo-controlled, Observer-blinded Phase 1 Study to Assess the Safety and Immunogenicity of Two Different Dose Levels of an Alum Adjuvanted Inactivated Whole Zika Virus Vaccine Candidate (VLA1601) in Healthy Flavivirus-naïve Adults Aged 18 to 49 Years
Brief Title: Randomized, Placebo-controlled, Observer-blinded Phase 1 Safety and Immunogenicity Study of Inactivated Zika Virus Vaccine Candidate in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Collaborators: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VLA1601-101
Record Dates: First submitted 2018-01-23; First posted 2018-02-07 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Zika Virus; Zika Virus Infection
Keywords: vaccine; prevention
MeSH Terms: conditions — Zika Virus Infection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: only dedicated site staff responsible for handling including preparation and administration of the vaccine will be unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment Group I (Experimental): 0.5 ml (6 antigen units (AU)) of VLA1601 on Day 0 and 28, 0.5 ml Placebo on Day 7
  Interventions: Biological: VLA1601; Biological: Placebo
- Treatment Group II (Experimental): 0.5 ml (6 antigen units (AU)) of VLA1601 on Day 0 and 7, 0.5 ml Placebo on Day 28
  Interventions: Biological: VLA1601; Biological: Placebo
- Treatment Group III (Experimental): 0.25 ml (3 antigen units (AU)) of VLA1601 on Day 0 and 28, 0.25 ml Placebo on Day 7
  Interventions: Biological: VLA1601; Biological: Placebo
- Treatment Group IV (Experimental): 0.25 ml (3 antigen units (AU)) of VLA1601 on Day 0 and 7, 0.25 ml Placebo on Day 28
  Interventions: Biological: VLA1601; Biological: Placebo
- Treatment Group V (Placebo Comparator): 0.5 ml Placebo on Day 0, 7 and 28
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VLA1601 — purified inactivated ZIKV vaccine candidate adsorbed on alum
  Arms: Treatment Group I; Treatment Group II; Treatment Group III; Treatment Group IV
Biological: Placebo — Phosphate buffered saline (PBS)

SUMMARY:
In this Phase 1 study, two target dose levels of VLA1601, a purified, inactivated, whole Zika virus (ZIKV) vaccine candidate adsorbed on aluminum hydroxide (alum) will be evaluated: 6 antigen units (AU) and 3 AU of inactivated ZIKV vaccine. Each dose will be administered intramuscularly (i.m.) in the deltoid muscle on Days 0 and 28. In addition, an accelerated 2-dose vaccination schedule on Days 0 and 7 will be assessed for both doses.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 to 49 years of age on the day of screening (Visit 0);
2. Subject has a Body Mass Index (BMI) of ≥18.5 and <30 kg/m2 on the day of screening (Visit 0);
3. Subject has an understanding of the study and its procedures, agrees to its provisions, and gives written informed consent prior to any study-related procedures;
4. Subject is generally healthy as determined by the Investigator's clinical judgment based on medical history, physical examination and screening laboratory tests;
5. If subject is of childbearing potential:

   i. Subject has a negative serum pregnancy test at screening (Visit 0);

ii. Subject agrees to employ adequate birth control measures for the duration of the study. This includes one of the following measures:

1. Hormonal contraceptives (e.g. implants, birth control pills, patches) since ≥30 days prior to first vaccination;
2. Intrauterine device;
3. Barrier type of birth control measure (e.g. condoms, diaphragms, cervical caps);
4. Vasectomy in the male sex partner ≥3 months prior to first vaccination;

Exclusion Criteria:

1. Subject has a history of known flavivirus infection, or vaccination with a licensed or investigational flavivirus vaccine;
2. Subject has plans to receive a licensed flavivirus vaccine during the course of the study;
3. Subject has plans to travel to areas (including within the US) with active ZIKV, Japanese Encephalitis Virus (JEV), Dengue Virus (DENV) or Yellow Fever Virus (YFV) transmission during the course of the study or has travelled to a flavivirus-endemic area within 4 weeks prior to study enrollment;
4. Subject is seropositive to ZIKV, JEV, DENV or West Nile virus (WNV);
5. Subject has received an inactivated vaccine within 2 weeks or live vaccine within 4 weeks prior to vaccination in this study;
6. Subject has clinically significant abnormal laboratory values, as determined by the Investigator, at screening (Visit 0);
7. Subject tests positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV);
8. Subject currently has or has a history of significant cardiovascular, respiratory (including asthma), metabolic, neurological (including Guillain-Barré syndrome), hepatic, rheumatic, autoimmune, hematological, gastrointestinal or renal disorder;
9. Subject has a disease or is undergoing a form of treatment or was undergoing a form of treatment within 4 weeks prior to study enrollment (i.e. subject randomized) that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (>800 μg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs (use of inhaled (low dose), intranasal or topical steroids is permitted);
10. Subject has a history of severe hypersensitivity reactions or anaphylaxis;
11. Subject has a history of any vaccine related contraindicating event (e.g., anaphylaxis, allergy to components of the candidate vaccine, other known contraindications);
12. Subject had acute febrile infections within two weeks prior to vaccination in this study;
13. Subject has donated blood within 30 days or received blood-derived products (e.g. plasma) within 90 days prior to vaccination in this study or plans to donate blood or use blood products during the course of the study;
14. Subject has a rash, dermatological condition or tattoos that would, in the opinion of the Investigator, interfere with injection site reaction rating;
15. Subject is currently enrolled or has participated in another clinical study involving an investigational medicinal product (IMP) or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an IMP or investigational device during the course of this study;
16. Subject has plans to become pregnant during the course of the study, or is pregnant (positive serum pregnancy test at screening) or lactating at the time of study enrollment;
17. Subject has a known or suspected problem with alcohol or drug abuse as determined by the Investigator;
18. Subject is committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities);
19. Subject is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the Investigator or site personnel conducting the study;
20. Subject has any condition that, in the opinion of the Investigator, may compromise the subject's well-being, might interfere with evaluation of study endpoints, or would limit the subject's ability to complete the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2018-02-24 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Rate of subjects with solicited adverse events including injection site and systemic reactions | within 7 days after any vaccination

SECONDARY OUTCOMES:
Rate of subjects with solicited adverse events including injection site and systemic reactions | within 7 days after each vaccination
Rate of subjects with any adverse events (AEs) | up to Day 56
Rate of subjects with any adverse events (AEs) | during the entire study period, i.e., up to Day 208
Rate of subjects with serious adverse events (SAEs) | up to Day 56
Rate of subjects with serious adverse events (SAEs) | up to Day 208
Rate of subjects with any IMP-related AEs | up to Day 56
  IMP: Investigational Medicinal Product;
Rate of subjects with any IMP-related AEs | up to Day 208
  IMP: Investigational Medicinal Product;
Rate of subjects with any IMP-related SAEs | up to Day 56
  IMP: Investigational Medicinal Product;
Rate of subjects with any IMP-related SAEs | up to Day 208
  IMP: Investigational Medicinal Product;
Geometric mean titer (GMT) for ZIKV-specific neutralizing antibody titer after last active vaccination | 7 days after last active vaccination
  GMT determined by plaque reduction neutralization test (PRNT)
Geometric mean titer (GMT) for ZIKV-specific neutralizing antibody titer after last active vaccination | 28 days after last active vaccination
  GMT determined by plaque reduction neutralization test (PRNT)
GMT for ZIKV-specific neutralizing antibody titer after first vaccination | 7 days after first vaccination
  GMT determined by PRNT
GMT for ZIKV-specific neutralizing antibody titer after first vaccination | 28 days after first vaccination
  for the Day 0, 28 schedule; GMT determined by PRNT
GMT for ZIKV-specific neutralizing antibody titer after first vaccination | Day 208 after first vaccination
  GMT determined by PRNT
Rate of subjects with seroconversion after last active vaccination | 7 days after last active vaccination
Rate of subjects with seroconversion after last active vaccination | 28 days after last active vaccination
Rate of subjects with seroconversion after first vaccination | 7 days after first vaccination
Rate of subjects with seroconversion after first vaccination | 28 days after first vaccination
  for the Day 0, 28 schedule
Rate of subjects with seroconversion after first vaccination | 208 days after first vaccination
Fold increase of ZIKV-specific neutralizing antibody titers after last active vaccination as compared to baseline | 7 after last active vaccination
Fold increase of ZIKV-specific neutralizing antibody titers after last active vaccination as compared to baseline | 28 after last active vaccination
Fold increase of ZIKV-specific neutralizing antibody titers after first vaccination as compared to baseline | 7 days after first vaccination
Fold increase of ZIKV-specific neutralizing antibody titers after first vaccination as compared to baseline | 28 days after first vaccination
  for the Day 0, 28 schedule
Fold increase of ZIKV-specific neutralizing antibody titers after first vaccination as compared to baseline | 208 days after first vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Dubischar, Study Director — Valneva Austria GmbH
Locations (1):
- New Orleans Center for Clinical Research, Knoxville, Tennessee, United States